CLINICAL TRIAL: NCT02392715
Title: Inspiratory Muscle Training Combined With General Exercise Training, Compared to General Exercise Training Alone in Patients With COPD: Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training Combined With General Exercise Training in COPD
Acronym: IMTGET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hôpital Riviera-Chablais, Vaud-Valais (Other)
Responsible Party: Principal Investigator, Stéphanie Vaudan, Stéphanie Vaudan, board-certified respiratory therapist, Hôpital Riviera-Chablais, Vaud-Valais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 003/15
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inspiratory muscle training; General exercise training; pulmonary rehabilitation; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention cohort (Experimental): 36 sessions of 60 - 75 minutes with a frequency of 3x/week
  30' endurance training, 15' strength training, 15' inspiratory muscle training with Threshold by Respironics
  Inspiratory muscle training intensity: 15% of maximal inspiratory pressure (PiMax) during the first week. Then increment of 5% each session until 60% of PiMax after the first month. The PiMax will be reassessed after 12 and 24 sessions in order to readjust the 60% of PiMax.
  Interventions: Device: Inspiratory muscle training with Threshold by respironics
- Control cohort (Sham Comparator): 36 sessions of 60 - 75 minutes with a frequency of 3x/week
  30' endurance training, 15' strength training, 15' sham inspiratory muscle training with Threshold by Respironics
  Sham inspiratory muscle training intensity : 5 centimeters of water (cmH20)
  Interventions: Device: Sham Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training with Threshold by respironics — Inspiratory muscle training
  15 minutes, 3x/weeks, 36 sessions
  Intensity: 15% of PiMax during the first week. Then increment of 5% each session until 60% of PiMax after the first month. The PiMax will be reassessed after 12 and 24 sessions in order to readjust the 60% of PiMax.
  Arms: Intervention cohort
Device: Sham Inspiratory muscle training — with Threshold by respironics
  15 minutes, 3x/weeks, 36 sessions
  Intensity: 5 centimeters of water (cmH20)
  Arms: Control cohort

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a frequent disease, with increasing prevalence. Pulmonary rehabilitation through general exercise training (GET) is a corner stone of COPD care. Inspiratory muscle training (IMT) as a stand-alone therapy decreases dyspnea and improves exercise capacity. Whether IMT combined with GET adds a supplementary benefit in the rehabilitation of COPD patients is however uncertain.

DETAILED DESCRIPTION:
Prospective, parallel-group, randomized controlled trial

80 COPD patients will be randomized into two groups. One group will receive general exercise training combined with inspiratory muscle training, 3 times a week, for a total of 36 sessions. The other group will receive general exercise training combined with shame inspiratory muscle training, 3 times a week, for a total of 36 sessions.

We will assess the difference of improvement in exercise capacity between the 2 groups with the 6 minute walking test. We will also assess the difference of improvement in quality of life with St-George's respiratory questionnaire. Finally the difference of improvement in maximal inspiratory pressure will be determined.

Patients and investigators assessing the outcomes will be blinded to group allocation.

Written informed consent will be obtained from each subject. The data will be treated anonymously.

ELIGIBILITY:
Inclusion Criteria:

* COPD demonstrated by spirometry using Gold Criteria
* Patient referred by a pneumologist to the ambulatory pulmonary rehabilitation program at the Riviera-Chablais Hospital, Monthey
* Patient with maximal inspiratory pressure < 60 cmH20
* Patient older than 40 years

Exclusion Criteria:

* Orthopaedic or neurological troubles that could slant the 6 minute walking test

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity (six minute walking test) | 12 weeks
  exercise capacity will be assessed by a six minute walking test

SECONDARY OUTCOMES:
Quality of Life (St-George's Respiratory questionnaire) | 12 weeks
  Quality of Life will be assessed by St-George's Respiratory questionnaire
Maximal inspiratory pressure (MicroRPM by MicroMedical) | 12 weeks
  Inspiratory maximal pressure will be assessed by the MicroRPM by MicroMedical

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Vaudan, BSc, Principal Investigator — stephanie.vaudan@hopitalrivierachablais.ch